CLINICAL TRIAL: NCT02121912
Title: Pilairo Q In-lab Market Research - Europe
Brief Title: Laboratory Assessment of Pilairo Q CPAP Mask Performance and Ease of Use.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CIA-89
Record Dates: First submitted 2014-04-14; First posted 2014-04-24 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-03

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- FPH Pilairo Q CPAP mask (Experimental): The Sleep Technician will fit the FPH Pilairo Q CPAP mask to the participant.
  Interventions: Device: FPH Pilairo Q CPAP mask
- Any other market released nasal or nasal-pillow CPAP mask (Active Comparator): The Sleep Technologist will fit the participant with any market released nasal or nasal-pillow CPAP mask
  Interventions: Device: Any other market released nasal or nasal-pillow CPAP mask

INTERVENTIONS:
Device: FPH Pilairo Q CPAP mask — CPAP nasal-pillow mask
  Other Names: FPH Pilairo CPAP mask; Pilairo Q; Pilairo
  Arms: FPH Pilairo Q CPAP mask
Device: Any other market released nasal or nasal-pillow CPAP mask — Any other market released nasal or nasal-pillow CPAP mask
  Arms: Any other market released nasal or nasal-pillow CPAP mask

SUMMARY:
Participants will undergo a normal sleep study. They will be randomised to use either a FPH Pilairo Q nasal pillow CPAP mask, or another mask. The sleep technician will record leak and pressure data, and complete questionnaires regarding satisfaction and ease of use at the end of the night. It is hypothesised that the Pilairo Q mask will be superior to other standard masks for CPAP therapy in terms of ease of use, satisfaction and overall titration experience.

DETAILED DESCRIPTION:
Participants will be recruited from patients who visit the sleep lab for CPAP titration. Only eligible participants, that provide written informed consent, will be enrolled into the investigation

Only those participants whom are previously diagnosed with an AHI >5 can be approached and enrolled into the study.

Once the consent form has been signed, participants will be randomly assigned to receive either Pilairo or any other standard care nasal/nasal pillows mask for their CPAP titration. A randomisation log will be provided by FPH.

The titration session will take place as per the lab's routine practice.

Throughout the night the Sleep Technician will record in the CRF the absolute leak value for the mask every 10 minutes.

At the end of the session the Sleep Technician will complete a questionnaire in relation to the titration experience for that participant/mask. The data will be collected in the CRF that FPH staff will provide to the site.

ELIGIBILITY:
Inclusion Criteria:

* AHI equal or greater than 15 from the diagnostic night.
* Equal or greater than 18 years of age

Exclusion Criteria:

* Inability to give informed consent.
* History of intolerance to CPAP.
* Anatomical or physiological conditions making CPAP therapy appropriate (for example a deviated septum)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martina Neddermann, Dr.med, Principal Investigator — Evangelisches Krankenhaus Herne
Locations (1):
- Evangelisches Krankenhaus Herne, Herne, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FPH Pilairo Q CPAP Mask | Any Other Market Released Nasal or Nasal-pillow CPAP Mask
Started | 25 | 25
Completed | 21 | 25
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FPH Pilairo Q CPAP Mask | Any Other Market Released Nasal or Nasal-pillow CPAP Mask | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Customized [Number; unit: participants] — Age information was only collected at the 18+ level. No other age information was collected.
  participants
    Age : 18 + years | 25 | 25 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 21 | 19 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Subjective Questionnaire of Mask Experience
Description: Sleep technicians reported on their experience using the mask after 1 night in the lab on a scale from 1 to 10 with a higher score indicating a better experience
Time Frame: 1 night in the lab
Population: While not all participants completed the full study, participants who provided acceptable data were used in the analysis. The number of participants analyzed may be different from the number who completed. Due to the nature of this study, participant completion did not have a direct effect on this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FPH Pilairo Q CPAP Mask | Any Other Market Released Nasal or Nasal-pillow CPAP Mask
Number analyzed (Participants) | 24 | 25
units on a scale | 8.08 (2.39) | 8.12 (2.37)

2. Secondary Outcome: Mask Leak
Description: The Sleep Technologist will record mask leak every 10minutes, over an 8 hour period during the sleep study.
Time Frame: Every 10min, for up to 8 hours
Measure: Mean (Standard Error); unit: liters/minute
Arm/Group | FPH Pilairo Q CPAP Mask | Any Other Market Released Nasal or Nasal-pillow CPAP Mask
Number analyzed (Participants) | 24 | 25
liters/minute | 38.36 (.99) | 35.47 (1.43)

3. Secondary Outcome: Sleep Technicians Recommendation to Use Mask
Description: Sleep Technicians reported on whether they would recommend the mask to other professionals. Ratings were out of 1-10 and a higher score indicates a higher likelihood of recommending the mask.
Time Frame: 1 night in the lab
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FPH Pilairo Q CPAP Mask | Any Other Market Released Nasal or Nasal-pillow CPAP Mask
Number analyzed (Participants) | 24 | 23
units on a scale | 8.83 (1.47) | 8.17 (1.85)

ADVERSE EVENTS:
Time Frame: 1 night 1 Night in Lab. Adverse event data was collected for the full time each participant remained in the trial, from informed consent until study completion or withdrawal. Each participant spent a different amount of time in the lab enrolled in the trial due to their sleep behavior. Therefore, a specific amount of time (or average) is not appropriate.
Arm/Group | FPH Pilairo Q CPAP Mask | Any Other Market Released Nasal or Nasal-pillow CPAP Mask
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 2/25 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FPH Pilairo Q CPAP Mask (N=25) | Any Other Market Released Nasal or Nasal-pillow CPAP Mask (N=25)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Low SpO2 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No